# Augmented Macular Pigment Supplement and Pericentral Visual Function: A Randomized Controlled Trial

NCT #: NCT04676126

Date: 28 April 2021

# Lumega-Z PLUS Randomized Controlled Trial Research Protocol

#### **Section 1: Purpose:**

The purpose of this study is to prospectively analyze changes in macular pigment ocular density and dermal carotenoid levels as they relate to perimetry in patients prescribed Lumega-Z, a medical food in combination with dorzolamide.

# **Section 2: Background and Significance:**

Macular pigments (MP) are a group of fat-soluble carotenoid polyenes that concentrate in the human macula and give it its characteristic yellow color. They are well studied compounds that optimize visual function and protect the macula from high energy visible light, inflammation, and oxidative damage.

Large historic randomized controlled trials have demonstrated that oral supplementation of lutein (L) and zeaxanthin (Z) are associated with macular protection and improvements in contrast sensitivity.<sup>3–5</sup> Recent investigations have demonstrated that the addition of the third macular pigment, meso-zeaxanthin (MZ) increases the bioavailability of both L and Z, and leads to higher MPOD than L and Z without MZ.<sup>6,7</sup>

Lumega-Z (LM) is a commercially available medical food that includes L, Z, and MZ, among other vitamins and minerals. Although this and other similar formulations have been shown to reduce risk of ARMD progression, the mechanisms of macular protection portend a benefit in other neurodegenerative processes as well. Indeed, high fidelity investigation of the effects of macular pigment supplements on memory has demonstrated measurable cognitive improvement.<sup>8</sup>

Glaucomatous neuron loss is a complex process with multiple contributing factors, and is not yet fully understood. Events that likely promote RGC apoptosis include disruption of neurotrophic factor axonal transport, It glutamate mediated excitotoxicity, It oxidative damage, It and autoimmune processes. It physical and chemical properties of the macular pigments suggest they act to attenuate the effects exerted by at least some of these mechanisms. The long polyene backbone of these carotenoids, for example, allows them to efficiently and sustainably dissipate energy from reactive oxygen species. Placeholds is a complex process with multiple contributing factors, and is not yet fully understood.

Two of the macular pigments, L and Z, are commonly found in the human diet, and blood levels respond directly to changes in dietary or supplemental intake. 17-19 Pressure mediated reflection spectroscopy has been shown to reliably measure dermal carotenoid levels, which correlate with plasma levels. This method can be used to non-invasively monitor carotenoid levels in glaucoma patients. 20-22

Dorzolamide is a topical carbonic anhydrase inhibitor (CAI) commonly used to treat glaucoma by inhibiting the production of aqueous humor to reduce intraocular pressure (IOP).<sup>23</sup> Incidentally, the targeted inhibition of carbonic anhydrase in the ocular circulation may have other effects on retinal and visual physiology, including increased retinal blood flow, improved perimetric light sensitivity, contrast sensitivity, and perimetric short wavelength sensitivity.<sup>24–26</sup> The vasodilation caused by topical CAI's suggest they may enhance delivery of the macular pigments to the retina, and so may have a synergistic benefit when paired with LM or other macular pigment-containing oral supplement.

Briefly, LM has demonstrated favorable effects on two objective measures of visual function: macular pigment optical density and contrast sensitivity, and an addition of a topical CAI may enhance delivery of the pigments to the macula. Anecdotal experience of the investigators suggests there may be an additional benefit in a subset of nutritionally vulnerable glaucoma patients. We therefore hypothesize that this subset of patients who experience improvement in visual field function after LM supplementation may be nutritionally or physiologically deficient of the macular pigments. This study will therefore prospectively examine the effects of LM supplementation in combination with a CAI on visual field function, MPOD, and CS in the context of a spectrophotometric analysis of dermal carotenoid levels in glaucoma patients compared to untreated controls.

# Section 3: Location, Facility and Equipment to Be Used:

#### LOCATION

311 Camden St, Ste 306, San Antonio, TX 78215

#### FACILITY

The medical office of Dr. William Sponsel

#### **EQUIPMENT**

- 1. Slit Lamp (Haag-Streit, Bern, Germany)
- 2. Veggie Meter (Longevity Link, Salt Lake City, Utah, USA)
- 3. MapcatSF (Guardion Health Sciences, San Diego, California, USA)
- 4. Vector Vision (Vector Vision Ocular Health, Greenville, Ohio, USA)
- 5. Humphrey Matrix Model 715 FDT Perimeter (Carl Zeiss Meditech, Jena, Germany)

# **Section 4: Subjects and Informed Consent**:

All subjects will be recruited from the medical practice of Dr. William E Sponsel. No advertising shall be employed. Eligible patients will be verbally informed of the study. If they express interest a detailed description of the study will be presented, including the written informed consent (attached) If they elect to participate, written informed consent will be obtained prior to any data collection. Consent documents will be available in both English and Spanish. Translation into Spanish will be performed by investigators fluent in the language. All study records will be anonymized and maintained on an encrypted and password protected computer under the control of the PI. Only aggregated mean results will be published in the scientific press.

## **PARTICIPANTS**

This prospective double-masked, randomized, placebo-controlled study will consist of 30 subjects age >18 with the diagnosis of Glaucoma (ICD-10: H40. \*). Only patients under the care of the investigating surgeon (WES) will be considered. Subjects will be identified at the time they are deemed to be candidates for Lumega-Z supplementation (adequate IOP control with RNFL or visual field glaucomatous progression). After verifying no history of AREDS formula oral supplement use, patients will be approached by the co-investigator (GTS) in the principal investigator's ophthalmology clinic and asked if they are interested in participating in this study. An Excel (Microsoft, Redmond, WA) spreadsheet with deidentified data will be kept in clinic on-site on a password-protected computer in

order to store and analyze data. GTS is a full-time employee at the investigating practice and has HIPPAA-compliant access to patients and patient records independent of this study.

#### INFORMED CONSENT

Before study participation, participants will have a consultation with a representative investigator at the clinical practice of WES (311 Camden St Ste. 306, San Antonio, TX, 78215) in which they will be informed of the risks, benefits, and alternatives of participating in the study. They will be assured that their decision to participate or not will have no bearing on their personal or medical treatment by the investigators. Subjects will be given a printed copy of their signed informed consent. Completed informed consent forms will be scanned and stored on their patient profile of a password protected and encrypted electronic medical record. After they are scanned onto the electronic medical record, the hard copies will be shredded. Participants will be given a copy of the signed informed consent forms.

#### **Inclusion Criteria**

- -Age ≥ 18 years
- -Glaucoma diagnosis (H40. \*) with abnormal visual field as measured by 30-2 Perimetry (mean deviation < -2.00)
- -Adequate IOP control (IOP > 7 mmHg and < 22 mmHg) by medical or surgical means measured by Goldman Applanation Tonometry for at least 3 months
- -Visual field progression decrease (more negative) in MD by 1.00 dB or more when compared to prior visual field)
- -Refractive error ≤ 10 diopters and astigmatism ≤ 3 diopters

## **Exclusion Criteria**

- -BCVA worse than 20/200
- -Pt Is unable to tolerate MPOD, CS, dermal carotenoid measurement-taking procedures
- -Patient reports taking LM supplement ≤ 2 times per week or cannot tolerate oral supplement intake
- -Patient loses IOP control and requires surgical intervention
- -Patient already taking AREDS formula oral supplement
- -Patient taking medication or dietary supplements that may interact with LM ingredients
- -History of photosensitive epilepsy
- -History of penetrating ocular trauma or vitrectomy
- -History of ocular or orbital radiation therapy or is currently receiving chemotherapy
- -Women who are nursing, pregnant, or are planning pregnancy
- -Has a known adverse reaction and/or sensitivity to the study supplement or its ingredients:

Including: N-acetyl-cysteine, acetyl-L-carnitine, L-taurine, quercetin, Co-enzyme Q-10, lutein, meso zeaxanthin, zeaxanthin, astazanthin, lycopene, alpha-lipoic acid.

- -Currently enrolled in an investigational drug study or has used an investigational drug within 30 days prior to recruitment.
- -Is planning on having ocular surgery at any time throughout the study duration, or had ocular surgery < 3 months before enrollment
- -Native lens opacity ≥ grade 3 on ARLNS standard photograph
- -Blue light filter intraocular lens
- -Sulfa Allergy

# **Section 5: Subject Compensation:**

Subjects will be compensated with gift cards according to the following schedule:

Visit 1: \$25

Visit 2: \$25

Visit 3: \$25

Visit 4: \$100

Funding will be provided by the study sponsor: Guardion Health Sciences, Inc.

## **Section 6: Duration:**

Patient recruitment, data collection, data analysis, and abstract/manuscript writing will take 6-12 months.

# Section 7: Research Design (Description of the Experiment, Data Collection and Analysis):

# 1. Study Design

This is a prospective double-masked, randomized controlled study which compares pre-Lumega-Z supplementation MPOD, CS, dermal carotenoid levels, and visual field status to post-supplement measurements of the same. Participants will be randomized to twelve weeks of LM + dorzolamide or twelve weeks of placebo. All packaging of LM and dorzolamide and their placebos will be identical and distributed by a third party. Both subjects and the investigators examining patients will be masked to placebo and experimental groups.

## 2. Supplement and CAI Dosing and Distribution

LumegaZ is a commercially available medical food (see ingredient table) which is consumed daily in a 1.5 Tbsp (0.75 FL OZ) dose. Subjects will be offered a 3-month supply (or placebo) for the duration of the study. Dosing instructions are included on the packaging.

The CAI which will be used in this study is Dorzolamide 2% ophthalmic solution used as follows: one drop in the affected (or both) eye three times per day. Dosing instructions are included on the packaging.

LumegaZ and CAI (or placebo) will be distributed upon recruitment in a single package which is identical to the standard LM supplement. Lot number will be recorded and used to determine whether subjects were in the placebo or supplement group after data gathering is complete.

| Ingredient | Amount | Ingredient | Amount |
|------------------|----------|--------------------|----------|
| Vitamin C | 500mg | Copper | 2 mg |
| Vitamin D3 | 2000 IU | Manganese | 2 mg |
| Vitamin E | 200 IU | Chromium | 120 mcg |
| Thiamin | 1.5mg | Molybdenum | 75 mcg |
| Riboflavin | 1.7mg | N-acetyl-cysteine | 500 mg |
| Vitamin B3 | 20 mg | Acetyl-L-Carnitine | 500 mg |
| Vitamin B6 | 10 mg | L-Taurine | 500 mg |
| Folate | 800mcg | Quercetin | 100 mg |
| Vitamin B12 | 1000 mcg | CoQ10 | 50 mg |
| Biotin | 100 mcg | Lutein | 15 mg |
| Panothenoic Acid | 10 mg | Meso-zeaxanthin | 3 mg |
| Calcium | 250 mg | Astaxanthin | 1000 mcg |
| Magnesium | 100 mg | Lycopene | 500 mcg |
| Zinc | 25 mg | Alpha-lipoic acid | 200mg |
| Selenium | 70 mcg | | |

#### 3. Randomization

After recruitment, subjects will be registered as a study participant and randomized by computer generated randomization table generated prior to subject recruitment to be in the placebo or intervention group by a Guardion Health Sciences representative without access to patient data. The Guardion representative will receive the subject name and delivery address only, which is the same information they receive for every patient prescribed this medical food.

The clinically active investigators and subjects will be masked to group assignment for the duration of the study. The placebo will be distributed directly to participants" homes in packaging identical to the standard LM product in a single shipment.

Dermal carotenoid measurement will be randomized by computer generated random number table to the right or left index finger of each subject at the initial visit. The same finger will be used at every follow-up visit.

MPOD is measured in one eye only, as there is very high correlation in values measured between eyes.<sup>27</sup> At the initial visit, the measured eye will be randomized by computer generated random number table. The same eye will be measured at every follow up visit.

# 4. Data Collection for dermal carotenoids, MPOD, and CS

All participants will have dermal carotenoid levels, MPOD, and CS measured at every visit up to 3 months after starting LM. The baseline measurements will be taken on the day of enrollment, then follow-up measurements will be taken 1 month, 2 months, and 3 months after initiation of topical dorzolamide + LM oral supplementation.

## a. Dermal Carotenoid Levels with Veggie Meter®

After finger randomization, the Veggie Meter® will be light- and dark- calibrated before every measurement. Smoking status, age, height, weight, handedness, and finger used will be documented at the time of data acquisition. Participants will be seated and insert the randomized index finger into the device, placed on a table at the level of the patients' heart. After a short wait of 3-10 seconds to allow for finger-tip compression by the device, optical data acquisition will begin (no blood sample is collected). After the ~5 seconds required to acquire data, the finger will be removed for ≥ 10 seconds to allow for recirculation of the tested finger. The measurement will be repeated 2 more times (for a total of 3 measurements per visit) and a carotenoid score will be reported and recorded as the average of the 3 values.

## b. Macular Pigment Optical Density with Heterochromatic Flicker Photometry

This data will be acquired as follows: After eye randomization the patient will be fitted into the device. They will be instructed to look at the center of a flashing circle and adjust the device to correct for their refractive error. A human operator will follow an independently developed algorithm (attached) to determine MPOD ± standard deviation, which will be calculated by the Mapcat device and recorded at each visit.

## c. Contrast Sensitivity with VectorVision

Participants will be asked to identify the location of a sine-wave gradient in a series of images by selecting the circle with the gradient as top, bottom, or neither. This will be repeated for all 4 different spatial frequencies and plotted on a contrast sensitivity curve.

## 5. Perimetry

All participants will have a baseline Frequency Doubling Technology (FDT) 10-2 taken no more than 1 month before starting LM supplementation. Follow-up FDT 10-2 testing will also be completed at 3 months after LM initiation.

#### 6. Power Analysis

The primary outcome measure in this study is dermal carotenoid levels, so power analysis with mean baseline score reported in the population is  $335 \pm 13.7$ , and conservative expected increase in carotenoid score to 360 with an alpha of 0.05 and a beta of 0.90 given a calculated n of 12 subjects. We will therefore recruit 30 subjects to participate in this study – 15 intervention and 15 controls.

## 7. Data Analysis

Pre-supplement dermal carotenoid scores, FDT 10-2 MD and pericentral sensitivity, MPOD, and CS parameters will be compared within subjects at the 1-month (except perimetry), 2-month (except perimetry), and 3-month time points using a two-way Repeated-measures ANOVA with post-hoc t-testing for evaluation of significant differences.

All investigators will contribute to data analysis.

## **Section 8: Risk Analysis:**

LM is a medical food with well-studied ingredients established to be safe, and are effective at preventing progression of mild-moderate age-related macular degeneration. A 10-year follow-up on the AREDS study cohort found zero MP-related adverse events in 4757 participants.<sup>28</sup>

Dorzolamide is a very common topical antiglaucoma medication. It is reasonably well tolerated, but adverse reactions may occur. These include ocular allergy, burning, stinging, and bitter taste. Burning and stinging may occur in as many as 40% of patients but this does not typically warrant discontinuation of the drug.<sup>29</sup> Preservative free formulations of dorzolamide can be used in cases of ocular allergy, and patients who cannot otherwise tolerate the stinging/burning will be excluded from the study.

MPOD tests involve looking at a flickering light. It is conceivable that in a predisposed individual, focusing on such a stimulus may trigger a seizure. <sup>30</sup> There are no reports in the literature of a Mapcat device triggering an epileptic seizure. As an added precaution, patients who are recruited for the study will be screened for a history of photosensitive seizures.

Dermal carotenoid measurement involves the application of moderate pressure on the index finger. This may cause pain in vulnerable patients, for example those with a history of arthritis or gout affecting the distal interphalangeal joint of the second digit. A physical exam by an investigating physician will identify patients who may be vulnerable to such pain and they will be informed that they can be removed from the study if they cannot tolerate the finger pressure.

Contrast sensitivity and involves identifying which of a set of circles has stripes. There are no known risks associated with conducting this test.

It is feasible that patients in the placebo group will be subject to increased risk of glaucomatous progression because they will not start on the topical carbonic anhydrase inhibitor, which has been shown to reduce IOP. Only patients with adequately controlled IOP will be included in the study, so topical CAI would otherwise not be indicated for their treatment regimen. Therefore, placebo patients

will still be receiving the standard of care for their glaucoma. Any patients with unexpected findings (such as elevated IOP) at any of the study visits requiring additional intervention will receive it.

#### **COVID-19 Statement**

The investigators acknowledge the current COVID-19 pandemic and associated risks. While the majority of COVID-19 infections are asymptomatic or mild severity, there is a risk of severe respiratory illness which can result in hospitalization, admission to the intensive care unit, intubation, chronic respiratory, cardiac, or neurologic sequalae, and death (risk varies widely and increases with age, although a global estimate is ~3%).<sup>31</sup>

Robust COVID-19 risk mitigation protocols are already in place at the investigating practice, which include the use of symptom and temperature screening, social distancing, intensive room and device cleaning with germicidal substances, thorough personal hygiene, use of personal protective equipment (PPE), and contact tracing and testing protocols to monitor exposed individuals. PPE includes N95 or equivalent facemasks, isolation gowns, gloves, eye protection, and plexiglass slit lamp face shields. Patients are also required to wear face masks at all times while in the clinic and are required to practice hand hygiene upon arrival. No patients with known or suspected COVID-19 infection are permitted in the clinic. These protocols are informed by, and exceed the requirements set forth by the US Centers for Disease Control.<sup>32</sup>

# **Section 9: Confidentiality:**

All records shall be anonymized and maintained on a password-protected encrypted computer under the control of the PI. Only aggregated, mean results will be published in the scientific press.

# **Section 10: Literature Cited:**

- 1. Bone RA, Landrum JT, Hime GW, Cains A, Zamor J. Stereochemistry of the human macular carotenoids. *Investig Ophthalmol Vis Sci.* Published online 1993.
- 2. Britton G. Structure and properties of carotenoids in relation to function. *FASEB J.* Published online 1995. doi:10.1096/fasebj.9.15.8529834
- 3. Chew EY, Clemons TE, SanGiovanni JP, et al. Secondary analyses of the effects of lutein/zeaxanthin on age-related macular degeneration progression AREDS2 report no. 3. *JAMA Ophthalmol*. Published online 2014. doi:10.1001/jamaophthalmol.2013.7376
- 4. Aronow ME, Chew EY. Age-related eye disease study 2: Perspectives, recommendations, and unanswered questions. *Curr Opin Ophthalmol*. Published online 2014. doi:10.1097/ICU.000000000000046
- 5. Akuffo KO, Beatty S, Peto T, et al. The impact of supplemental antioxidants on visual function in nonadvanced age-related macular degeneration: A head-to-head randomized clinical trial. *Investig Ophthalmol Vis Sci.* Published online 2017. doi:10.1167/iovs.16-21192
- 6. Bone RA, Davey PG, Roman BO, Evans DW. Efficacy of commercially available nutritional supplements: Analysis of serum uptake, macular pigment optical density and visual functional response. *Nutrients*. Published online 2020. doi:10.3390/nu12051321
- 7. Ma L, Liu R, Du JH, Liu T, Wu SS, Liu XH. Lutein, zeaxanthin and meso-zeaxanthin supplementation associated with macular pigment optical density. *Nutrients*. Published online 2016. doi:10.3390/nu8070426
- 8. Power R, Coen RF, Beatty S, et al. Supplemental Retinal Carotenoids Enhance Memory in Healthy

- Individuals with Low Levels of Macular Pigment in A Randomized, Double-Blind, Placebo-Controlled Clinical Trial. *J Alzheimer's Dis*. Published online 2018. doi:10.3233/JAD-170713
- 9. Almasieh M, Wilson AM, Morquette B, Cueva Vargas JL, Di Polo A. The molecular basis of retinal ganglion cell death in glaucoma. *Prog Retin Eye Res*. Published online 2012. doi:10.1016/j.preteyeres.2011.11.002
- 10. Quigley HA. Glaucoma. In: *The Lancet*.; 2011. doi:10.1016/S0140-6736(10)61423-7
- 11. Knox DL, Eagle RC, Green WR. Optic nerve hydropic axonal degeneration and blocked retrograde axoplasmic transport: Histopathologic features in human high-pressure secondary glaucoma. *Arch Ophthalmol*. Published online 2007. doi:10.1001/archopht.125.3.347
- 12. Tsai T, Reinehr S, Maliha AM, Joachim SC. Immune Mediated Degeneration and Possible Protection in Glaucoma. *Front Neurosci*. Published online 2019. doi:10.3389/fnins.2019.00931
- 13. Pinazo-Durán MD, Zanón-Moreno V, Gallego-Pinazo R, García-Medina JJ. Oxidative stress and mitochondrial failure in the pathogenesis of glaucoma neurodegeneration. In: *Progress in Brain Research*.; 2015. doi:10.1016/bs.pbr.2015.06.001
- 14. Greco A, Rizzo MI, De Virgilio A, Gallo A, Fusconi M, de Vincentiis M. Emerging Concepts in Glaucoma and Review of the Literature. *Am J Med*. Published online 2016. doi:10.1016/j.amjmed.2016.03.038
- 15. Wax MB. The case for autoimmunity in glaucoma. *Exp Eye Res*. Published online 2011. doi:10.1016/j.exer.2010.08.016
- 16. Foote CS, Chang YC, Denny RW. Chemistry of Singlet Oxygen. X. Carotenoid Quenching Parallels Biological Protection. *J Am Chem Soc.* Published online 1970. doi:10.1021/ja00720a036
- 17. Jahns L, Johnson LAK, Mayne ST, et al. Skin and plasma carotenoid response to a provided intervention diet high in vegetables and fruit: Uptake and depletion kinetics. *Am J Clin Nutr*. Published online 2014. doi:10.3945/ajcn.114.086900
- 18. Jahns L, Johnson LAK, Conrad Z, et al. Concurrent validity of skin carotenoid status as a concentration biomarker of vegetable and fruit intake compared to multiple 24-h recalls and plasma carotenoid concentrations across one year: a cohort study. *Nutr J*. Published online 2019. doi:10.1186/s12937-019-0500-0
- 19. Conrady CD, Bell JP, Besch BM, et al. Correlations between macular, skin, and serum carotenoids. *Investig Ophthalmol Vis Sci.* Published online 2017. doi:10.1167/iovs.17-21818
- 20. Ermakov I V., Gellermann W. Dermal carotenoid measurements via pressure mediated reflection spectroscopy. *J Biophotonics*. Published online 2012. doi:10.1002/jbio.201100122
- 21. Mayne ST, Cartmel B, Scarmo S, Jahns L, Ermakov I V., Gellermann W. Resonance Raman spectroscopic evaluation of skin carotenoids as a biomarker of carotenoid status for human studies. *Arch Biochem Biophys*. Published online 2013. doi:10.1016/j.abb.2013.06.007
- 22. Obana A, Tanito M, Gohto Y, Okazaki S, Gellermann W, Bernstein PS. Changes in macular pigment optical density and serum lutein concentration in Japanese subjects taking two different lutein supplements. *PLoS One*. Published online 2015. doi:10.1371/journal.pone.0139257
- 23. Schmidl D, Schmetterer L, Garhöfer G, Popa-Cherecheanu A. Pharmacotherapy of Glaucoma. *J Ocul Pharmacol Ther*. Published online 2015. doi:10.1089/jop.2014.0067
- 24. Stefánsson E, Pedersen DB, Jensen PK, et al. Optic nerve oxygenation. *Prog Retin Eye Res*. Published online 2005. doi:10.1016/j.preteyeres.2004.09.001
- 25. Sponsel WE, Harrison J, Elliott WR, Trigo Y, Kavanagh J, Harris A. Dorzolamide hydrochloride and visual function in normal eyes. *Am J Ophthalmol*. Published online 1997. doi:10.1016/S0002-9394(14)71124-9
- 26. Remky A, Weber A, Arend O, Sponsel WE. Topical dorzolamide increases pericentral visual function in age-related maculopathy: Pilot study findings with short-wavelength automated perimetry. *Acta Ophthalmol Scand*. Published online 2005. doi:10.1111/j.1600-

- 0420.2005.00406.x
- 27. Hammond BR, Fuld K. Interocular differences in macular pigment density. *Investig Ophthalmol Vis Sci.* Published online 1992.
- 28. Chew EY, Clemons TE, Agrón E, et al. Long-term effects of vitamins C and E, β-carotene, and zinc on age-related macular degeneration: AREDS Report No. 35. *Ophthalmology*. Published online 2013. doi:10.1016/j.ophtha.2013.01.021
- 29. Katz LJ, Simmons ST, Craven ER. Efficacy and safety of brimonidine and dorzolamide for intraocular pressure lowering in glaucoma and ocular hypertension. *Curr Med Res Opin*. Published online 2007. doi:10.1185/030079907X242476
- 30. Padmanaban V, Inati S, Ksendzovsky A, Zaghloul K. Clinical advances in photosensitive epilepsy. *Brain Res.* Published online 2019. doi:10.1016/j.brainres.2018.07.025
- 31. Ortiz-Prado E, Simbaña-Rivera K, Gómez- Barreno L, et al. Clinical, molecular, and epidemiological characterization of the SARS-CoV-2 virus and the Coronavirus Disease 2019 (COVID-19), a comprehensive literature review. *Diagn Microbiol Infect Dis*. Published online 2020. doi:10.1016/j.diagmicrobio.2020.115094
- 32. US Centers for Disease Control and Prevention. Interim Infection Prevention and Control Recommendations for Healthcare Personnel During the Coronavirus Disease 2019 (COVID-19) Pandemic. Accessed September 18, 2020. https://www.cdc.gov/coronavirus/2019-ncov/hcp/infection-control-recommendations.html